CLINICAL TRIAL: NCT04021511
Title: Early Prescription of Radiography Using the Ottawa Ankle Rules by a Nurse in the Management of Isolated Ankle Trauma at the Emergency Department's Reception of the Hospital Center of Saint-Brieuc
Brief Title: Early Prescription of Radiography Using the Ottawa Ankle Rules by a Nurse in the Management of Isolated Ankle Trauma
Acronym: PARIAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Saint-Brieuc (Other)
Responsible Party: Principal Investigator, Pierre Kergaravat, Hospital physician, principal Investigator, Centre Hospitalier de Saint-Brieuc
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CHSB_201905_P1_PARIAO
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Ankle Injuries; Nurse's Role; Emergencies
Keywords: overcrowding; x rays; emergency department; Ottawa Ankle Rules; nurse practitioner
MeSH Terms: conditions — Ankle Injuries; Emergencies; Crowding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase A (No Intervention): The first one (Phase A) will occur in the emergency department with the application of OAR only by the physicians (without changing the standard of care) during 4 weeks
- Phase B (Experimental): The second one (Phase B) will occur after the Phase A. Nurses will apply OAR according to the protocol. This phase will also lasts 4 weeks.
  Interventions: Other: OAR application by a nurse

INTERVENTIONS:
Other: OAR application by a nurse — As per protocol, in the Phase B, nurses will be allowed to apply OAR which can lead to an early radiography prescription.
  Arms: Phase B

SUMMARY:
The study will be conducted in 2 phases (A and B) using two different groups of patients in order to prove that an early prescription of radiography using the Ottawa Ankle Rules by a nurse practitioner could shorten length of stay of a patient suffering from ankle trauma at the Hospital Center of Saint-Brieuc.

DETAILED DESCRIPTION:
Ankle sprain is an injury very frequently encountered during consultation in hospitals emergency departments. Its mechanism may at times leads to fracture. The Ottawa Ankle Rules (OAR) provide guidelines to clinicians concerning the need to perform radiographic test to verify whether patients with ankle injuries are suffering from fracture. If all clinical and anamnestic criteria are negative in accordance with the OAR, the probability of a fracture being present is about 0% (IC 95%). OAR are validated for adults.

Actually, a meta-analysis has suggested that it may be beneficial to introduce a nurse-initiated radiographic test protocol as a standard practice in emergency departments. However this early prescription is not a standard of care in most of emergency departments in France.

The implementation of OAR decreases irradiation levels of patients and reduces medical expenses. In addition, it allows to reduce patient's duration of stay in already encumbered emergency departments, thus reducing also overcrowding, which is known to be a major factor of non quality of care in such departments.

The study will be conducted in 2 phases of 4 weeks each :

* The first one (Phase A) will occur in the emergency department with the application of OAR only by the physicians (without changing the standard of care)
* The second one (Phase B) will occur after the Phase A, and nurses will apply OAR before physicians, according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* With closed ankle injury less than 10 days old
* Affiliation to the national health insurance
* Written informed consent must be obtained

Exclusion Criteria:

* Trauma dating more than 10 days
* Patient not affiliated to the national health insurance
* X-ray performed before patient admission
* Other trauma than an isolated trauma of the ankle
* Injury other than ankle injury : calcaneus, toes, and Achilles' tendon
* Paraplegic or quadriplegic patient
* Previous admission to the Emergency Department for the same traumatic event
* Patient already included in the PARIAO study
* Isolated skin injury / isolated superficial injury
* Ankle fracture or obvious deformation
* Neuro-vascular deficit
* Mental disorder
* Adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty
* Excessive alcoholization or intoxication by other psychoactive substances (physician's decision)
* Uncooperative patient
* Pregnancy in progress

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Time spent in emergency departement | through study completion, between 2 and 3 months
  Difference of time spent in minutes in emergency department between Phase A group and Phase B group.

SECONDARY OUTCOMES:
Percentage of x-rays | through study completion, between 2 and 3 months
  Difference of the percentage of x-rays between Phase A group and Phase B group.
Time spent by nurse for patient care | through study completion, between 2 and 3 months
  Difference of the time spent by nurse for patient care between Phase A group and Phase B group.
Comparaison of x-rays prescription between physicians and nurses | through study completion, between 2 and 3 months
  Difference of percentage of x-rays prescribed by nurses and physicians in Phase B group.
Numbers of fractures identified by an x-ray requested by the physician in group B | through study completion, between 2 and 3 months
  For patients who have a fracture identified by an x-ray requested by the nurse or the physician : number of X-rays not requested by the nurse in the Phase B group.
Numbers of fractures identified by an x-ray requested by a nurse in group B | through study completion, between 2 and 3 months
  For patients who have a fracture identified by an x-ray requested by the nurse or the physician : number of X-rays not requested by the physician.
Other x-rays required | through study completion, between 2 and 3 months
  For patients whose x-ray was required, percentage of ankle x-ray performed while actually the trauma concerned the foot and not the ankle.
Satisfaction rate of nurses | through study completion, between 2 and 3 months
  Satisfaction rate of nurses evaluated through a questionnaire with 5 questions.
  Tittle : Nurse's satisfaction survey
  1. - evaluation of nurse's satisfaction for management of ankle trauma in usual management : scale from 0 to 10. 0 is no satisfaction ; 10 is important satisfaction.
  2. - evaluation of nurse's satisfaction for management of ankle trauma in this new management : scale from 0 to 10. 0 is no satisfaction ; 10 is important satisfaction.
  3. - question about Ottawa Ankle Rules application : does nurse think that this rules application improves patient's management (quality, quickness, …) ? : yes or no
  4. - evaluation of additional workload for nurse with the new management : scale from 0 to 10. 0 is no additional workload ; 10 is important additional workload
  5. - question if nurse is ready from now to realize an early prescription of radiography using the Ottawa Ankle Rules : yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Brieuc, Saint-Brieuc, France

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data (anonymized) that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: From the end of the study for 15 years.
Access Criteria: Access through secure platform with personal username and password

REFERENCES:
- [Result] Stiell IG, Greenberg GH, McKnight RD, Nair RC, McDowell I, Worthington JR. A study to develop clinical decision rules for the use of radiography in acute ankle injuries. Ann Emerg Med. 1992 Apr;21(4):384-90. doi: 10.1016/s0196-0644(05)82656-3. PMID 1554175
- [Result] Stiell IG, Greenberg GH, McKnight RD, Nair RC, McDowell I, Reardon M, Stewart JP, Maloney J. Decision rules for the use of radiography in acute ankle injuries. Refinement and prospective validation. JAMA. 1993 Mar 3;269(9):1127-32. doi: 10.1001/jama.269.9.1127. PMID 8433468
- [Result] Stiell I, Wells G, Laupacis A, Brison R, Verbeek R, Vandemheen K, Naylor CD. Multicentre trial to introduce the Ottawa ankle rules for use of radiography in acute ankle injuries. Multicentre Ankle Rule Study Group. BMJ. 1995 Sep 2;311(7005):594-7. doi: 10.1136/bmj.311.7005.594. PMID 7663253
- [Result] Fan J, Woolfrey K. The effect of triage-applied Ottawa Ankle Rules on the length of stay in a Canadian urgent care department: a randomized controlled trial. Acad Emerg Med. 2006 Feb;13(2):153-7. doi: 10.1197/j.aem.2005.07.041. Epub 2006 Jan 25. PMID 16436790
- [Result] Ho JK, Chau JP, Cheung NM. Effectiveness of emergency nurses' use of the Ottawa Ankle Rules to initiate radiographic tests on improving healthcare outcomes for patients with ankle injuries: A systematic review. Int J Nurs Stud. 2016 Nov;63:37-47. doi: 10.1016/j.ijnurstu.2016.08.016. Epub 2016 Aug 25. PMID 27592083
- [Result] Allerston J, Justham D. Nurse practitioners and the Ottawa Ankle Rules: comparisons with medical staff in requesting X-rays for ankle injured patients. Accid Emerg Nurs. 2000 Apr;8(2):110-5. doi: 10.1054/aaen.2000.0103. PMID 10818378
- [Result] Derlet RW, Richards JR. Overcrowding in the nation's emergency departments: complex causes and disturbing effects. Ann Emerg Med. 2000 Jan;35(1):63-8. doi: 10.1016/s0196-0644(00)70105-3. PMID 10613941
- [Result] Lau LH, Kerr D, Law I, Ritchie P. Nurse practitioners treating ankle and foot injuries using the Ottawa Ankle Rules: a comparative study in the emergency department. Australas Emerg Nurs J. 2013 Aug;16(3):110-5. doi: 10.1016/j.aenj.2013.05.007. Epub 2013 Jun 25. PMID 23953094